CLINICAL TRIAL: NCT00488059
Title: A Multicenter, Open-label Study Evaluating the Antiviral Activity and Safety of Enfuvirtide (ENF) Once Daily (QD) or Twice Daily (BID) in Triple-class Experienced HIV-1 Infected Patients Changing Their Therapy to a Standard of Care (SOC) Regimen That Includes Initiating Raltegravir Plus an Optimized Background (OB) Antiviral Regimen
Brief Title: A Study of Fuzeon (Enfuvirtide) With an Integrase Inhibitor Plus Optimized Background in Treatment-Experienced HIV-1 Infected Patients
Acronym: AMICI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was terminated early due to poor enrollment.
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Trimeris (Industry)
Responsible Party: Clinical Trials, Study Director, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20837
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Results first posted 2011-06-29 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide; Integrase Inhibitors

ARMS (2):
- Phase I (Experimental): Phase 1: ENF 90mg SC BID): In the first phase or cohort phase of day I-1 through Week I-12 of the trial all patients received enfuvirtide (ENF) 90 mg subcutaneously (SC) twice daily (BID) + Isentress® [raltegravir] (RAL) 400-mg orally (PO) BID + optimized background (OB) with at least 1 fully active antiretroviral (ARV) agent excluding nucleoside reverse transcriptase inhibitor (NRTIs).
  Interventions: Drug: enfuvirtide [Fuzeon]; Drug: Optimized background ARV; Drug: Integrase inhibitor
- Phase II (Experimental): In the randomized comparator Phase II of the trial- (Day II-1 through Week II-16): Virologic responders confirmed HIV-1 RNA ≤50 copies/mL from Phase I were randomized to 1 of 2 treatment arms of
  (Phase II Arm A: Phase I then ENF 90mg SC BID): ENF 90 mg SC BID + RAL 400 mg PO BID + OB with at least 1 fully active ARV agent excluding NRTIs or (Phase II Arm B: Phase I then ENF 180mg SC QD): ENF 180 mg SC once daily (QD) + RAL 400 mg PO BID + OB with at least 1 fully active ARV agent excluding NRTIs.
  Interventions: Drug: Optimized background ARV; Drug: Integrase inhibitor; Drug: enfuvirtide [Fuzeon]

INTERVENTIONS:
Drug: enfuvirtide [Fuzeon] — 90 mg SC twice daily
  Arms: Phase I
Drug: Optimized background ARV — As prescribed
Drug: Integrase inhibitor — As prescribed
Drug: enfuvirtide [Fuzeon] — 180 mg SC once daily
  Arms: Phase II

SUMMARY:
This 2-arm study evaluated the efficacy and safety of Fuzeon with an integrase inhibitor in an expanded access program plus an optimized background antiviral regimen (AVR) in HIV-1 infected patients naive to Fuzeon and an integrase inhibitor. In the first cohort phase of the study (Phase I), eligible patients received Fuzeon 90 mg subcutaneously (SC) twice daily until confirmation of response (min/max = 8/16 weeks). In Phase II, the randomised comparator phase of the study, responders were randomized to receive Fuzeon either 90 mg SC twice a day or 180 mg SC once a day for a further 16 weeks. Non-responders and virological failures were terminated from the study. The anticipated time on study treatment was 3-9 months, and the target sample size was 210 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >=18 years of age
* HIV-1 infection
* Triple class treatment-experienced, Fuzeon- and integrase-inhibitor naive
* GSS >= 3 ; nucleosides excluded

Exclusion Criteria:

* Adverse clinical or laboratory experience >ACTG Grade 4
* Untreated infection, intercurrent illness, drug toxicity or other condition contraindicating an antiretroviral regimen
* Malignancy requiring chemotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United States (36):
  - Hobson City, Alabama
  - Phoenix, Arizona
  - Los Angeles, California
  - Modesto, California
  - Stanford, California
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - North Palm Beach, Florida
  - Orlando, Florida
  - Plantation, Florida
  - Port Saint Lucie, Florida
  - Safety Harbor, Florida
  - South Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Silver Spring, Maryland
  - Boston, Massachusetts
  - Kansas City, Missouri
  - St Louis, Missouri
  - Newark, New Jersey
  - Briarcliff Manor, New York
  - New York, New York
  - Rochester, New York
  - The Bronx, New York
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Reading, Pennsylvania
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Annandale, Virginia
- Puerto Rico (2):
  - Ponce
  - Santurce

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase I of the study was a single group. In Phase II of the study, the remaining patients were randomized to either the enfuvirtide (90 mg) BID group or the enfuvirtide (180 mg) QD group.
Groups:
- Phase I: (Phase 1: ENF 90mg SC BID): In the first phase or cohort phase of day I-1 through Week I-12 of the trial all patients received enfuvirtide (ENF) 90 mg subcutaneously (SC) twice daily (BID) + Isentress® [raltegravir] (RAL) 400-mg orally (PO) BID + optimized background (OB) with at least 1 fully active antiretroviral (ARV) agent excluding nucleoside reverse transcriptase inhibitor (NRTIs).
- Phase II - Arm A: Phase I then enfuvirtide 90 mg SC BID + RAL 400 mg PO BID + OB (with at least 1 fully active ARV agent excluding NRTIs)
- Phase II - Arm B: Phase I then enfuvirtide 180 mg SC QD (2 x 90-mg injections) + RAL 400 mg PO BID + OB (with at least 1 fully active ARV agent excluding NRTIs)
Period: Phase I: ENF 90mg SC BID
Arm/Group | Phase I | Phase II - Arm A | Phase II - Arm B
Started | 29 | 0 | 0
Completed | 14 | 0 | 0
Not Completed | 15 | 0 | 0
Period: Phase II Arm A:Phase I Then ENF 90mg BID
Arm/Group | Phase I | Phase II - Arm A | Phase II - Arm B
Started | 0 | 9 | 0
Completed | 0 | 7 | 0
Not Completed | 0 | 2 | 0
Period: Phase II Arm B:Phase I Then ENF 180mg QD
Arm/Group | Phase I | Phase II - Arm A | Phase II - Arm B
Started | 0 | 0 | 5
Completed | 0 | 0 | 1
Not Completed | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: ENF 90mg SC BID: (Phase 1: ENF 90mg SC BID): In the first phase or cohort phase of day I-1 through Week I-12 of the trial all patients received enfuvirtide (ENF) 90 mg subcutaneously (SC) twice daily (BID) + Isentress® [raltegravir] (RAL) 400-mg orally (PO) BID + optimized background (OB) with at least 1 fully active antiretroviral (ARV) agent excluding nucleoside reverse transcriptase inhibitor (NRTIs).
Arm/Group | Phase 1: ENF 90mg SC BID
Number analyzed (Participants) | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 45.4 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Phase I of the Study With a Confirmed HIV-1 RNA Viral Load ≤ 50 Copies/mL
Description: Virologic responders were defined as patients who had an initial HIV-1 RNA assessment <= 50 copies/mL during Phase I at any visit between Week I-4 and Week I-12 and a confirmatory viral load assessment ≤ 50 copies/mL at the next visit (Week I-8 to Week II-16)
Time Frame: Between Week I-4 and Week I-12 of Phase I of the study
Population: Intent-to-treat population
Measure: Number; unit: participants
Groups:
- Phase I: ENF 90mg SC BID: (Phase 1: ENF 90mg SC BID): In the first phase or cohort phase of day I-1 through Week I-12 of the trial all patients received enfuvirtide (ENF) 90 mg subcutaneously (SC) twice daily (BID) + Isentress® [raltegravir] (RAL) 400-mg orally (PO) BID + optimized background (OB) with at least 1 fully active antiretroviral (ARV) agent excluding nucleoside reverse transcriptase inhibitor (NRTIs).
Arm/Group | Phase I: ENF 90mg SC BID
Number analyzed (Participants) | 29
participants
  Week 8 | 8
  Week 12 | 5
  Week 16 | 1

2. Secondary Outcome: Virologic Response Over Time in Phase I of the Study
Description: The number of intent-to-treat (ITT) participants with HIV-1 RNA <= 50 copies/mL and HIV-1 RNA < 400 copies/mL by study week are summarized below.
Time Frame: Weeks 4, 8 & 12
Population: Intent-to-treat population
Measure: Number; unit: participants
Arm/Group | Phase I: ENF 90mg SC BID
Number analyzed (Participants) | 29
participants
  Week 4 (<= 50 copies/mL) | 11
  Week 4 (< 400 copies/mL) | 22
  Week 8 (<= 50 copies/mL) | 14
  Week 8 (< 400 copies/mL) | 22
  Week 12 (<= 50 copies/mL) | 14
  Week 12 (< 400 copies/mL) | 19

3. Primary Outcome: Number of Patients in Phase II of the Study With HIV-1 RNA ≤ 50 Copies/mL at Week II-16
Time Frame: Week II-16
Population: Intent-to-treat population
Measure: Number; unit: participants
Groups:
- Phase II Arm A: Phase I Then ENF 90 mg SC BID: (Phase 1: ENF 90 mg SC BID): In the first phase or cohort phase of day I-1 through Week I-12 of the trial all patients received enfuvirtide (ENF) 90 mg subcutaneously (SC) twice daily (BID) + Isentress® [raltegravir] (RAL) 400-mg orally (PO) BID + optimized background (OB) with at least 1 fully active antiretroviral (ARV) agent excluding nucleoside reverse transcriptase inhibitor (NRTIs).
  In the randomized comparator phase Phase II of the trial- (Day II-1 through Week II-16): Virologic responders confirmed HIV-1 RNA ≤50 copies/mL)from Phase I were randomized to
  (Phase II Arm A: Phase I+ENF 90mg SC BID): ENF 90 mg SC BID + RAL 400 mg PO BID + OB with at least 1 fully active ARV agent excluding NRTIs.
- Phase II Arm B: Phase I Then ENF 180mg SC QD: (Phase 1: ENF 90 mg SC BID): In the first phase or cohort phase of day I-1 through Week I-12 of the trial all patients received enfuvirtide (ENF) 90 mg subcutaneously (SC) twice daily (BID) + Isentress® [raltegravir] (RAL) 400-mg orally (PO) BID + optimized background (OB) with at least 1 fully active antiretroviral (ARV) agent excluding nucleoside reverse transcriptase inhibitor (NRTIs).
  In the randomized comparator phase Phase II of the trial- (Day II-1 through Week II-16): Virologic responders confirmed HIV-1 RNA ≤50 copies/mL)from Phase I were randomized to
  (Phase II Arm B: Phase I then ENF 180mg SC QD): ENF 180 mg SC once daily (QD) + RAL 400 mg PO BID + OB with at least 1 fully active ARV agent excluding NRTIs.
Arm/Group | Phase II Arm A: Phase I Then ENF 90 mg SC BID | Phase II Arm B: Phase I Then ENF 180mg SC QD
Number analyzed (Participants) | 9 | 5
participants | 5 | 3

4. Secondary Outcome: HIV-1 RNA Viral Load Change From Baseline in Phase I of the Study
Description: Change from baseline in HIV-1 RNA (log10 copies/mL) at study Weeks I-4, 8, 12 & LOCF for ITT patients in Phase I of the study
Time Frame: Baseline and Weeks 4, 8, 12 & LOCF
Population: Intent-to-treat population. Last Observation Carried Forward (LOCF) includes non-missing data values from the last post-baseline visit for each participant which was carried forward to impute missing data values.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Phase I: ENF 90mg SC BID
Number analyzed (Participants) | 29
log10 copies/mL
  Baseline (N=29) | 4.4 (0.87)
  change at Week 4 (n=27) | 2.1 (0.46)
  change at Week 8 (n=24) | 2.0 (0.81)
  change at Week 12 (n=14) | 2.4 (1.09)
  change at Week 16 (n=10) | 2.3 (0.90)
  change at LOCF (n=27) | 1.9 (0.61)

5. Secondary Outcome: Virologic Response Over Time in Phase II of the Study
Description: The number of intent-to-treat (ITT) participants with HIV-1 RNA <= 50 copies/mL and HIV-1 RNA < 400 copies/mL by study week.
Time Frame: Weeks II-4, 8, 12 & 16
Population: intent-to-treat population
Measure: Number; unit: participants
Groups:
- Phase II Arm A: Phase I Then ENF 90mg SC BID: (Phase 1: ENF 90 mg SC BID): In the first phase or cohort phase of day I-1 through Week I-12 of the trial all patients received enfuvirtide (ENF) 90 mg subcutaneously (SC) twice daily (BID) + Isentress® [raltegravir] (RAL) 400-mg orally (PO) BID + optimized background (OB) with at least 1 fully active antiretroviral (ARV) agent excluding nucleoside reverse transcriptase inhibitor (NRTIs).
  In the randomized comparator phase Phase II of the trial- (Day II-1 through Week II-16): Virologic responders confirmed HIV-1 RNA ≤50 copies/mL)from Phase I were randomized to
  (Phase II Arm A: Phase I then ENF 90mg SC BID): ENF 90 mg SC BID + RAL 400 mg PO BID + OB with at least 1 fully active ARV agent excluding NRTIs.
Arm/Group | Phase II Arm A: Phase I Then ENF 90mg SC BID | Phase II Arm B: Phase I Then ENF 180mg SC QD
Number analyzed (Participants) | 9 | 5
participants
  Week 4 (<= 50 copies/mL) | 5 | 4
  Week 4 (< 400 copies/mL) | 6 | 4
  Week 8 (<= 50 copies/mL) | 6 | 4
  Week 8 (< 400 copies/mL) | 7 | 4
  Week 12 (<= 50 copies/mL) | 6 | 4
  Week 12 (< 400 copies/mL) | 7 | 4
  Week 16 (<= 50 copies/mL) | 5 | 3
  Week 16 (< 400 copies/mL) | 6 | 4

6. Secondary Outcome: CD4+ Lymphocyte Count Change From Baseline
Description: Change from study Phase I baseline in CD4+ lymphocyte count at Phase II study Weeks II - 1, 12, 16, and LOCF by treatment arm.
  Change from study Phase II baseline in CD4+ lymphocyte count at Phase II study weeks II - 12 and 16.
Time Frame: Phase I Baseline and Phase II Weeks II-1, 12, 16, and LOCF
Population: Intent-to-treat
Measure: Median (Full Range); unit: cells/mm3
Groups:
- Phase II Arm A: Phase I Then ENF 90mg BID: (Phase 1: ENF 90 mg SC BID): In the first phase or cohort phase of day I-1 through Week I-12 of the trial all patients received enfuvirtide (ENF) 90 mg subcutaneously (SC) twice daily (BID) + Isentress® [raltegravir] (RAL) 400-mg orally (PO) BID + optimized background (OB) with at least 1 fully active antiretroviral (ARV) agent excluding nucleoside reverse transcriptase inhibitor (NRTIs).
  In the randomized comparator phase Phase II of the trial- (Day II-1 through Week II-16): Virologic responders confirmed HIV-1 RNA ≤50 copies/mL)from Phase I were randomized to
  (Phase II Arm A: Phase I then ENF 90mg SC BID): ENF 90 mg SC BID + RAL 400 mg PO BID + OB with at least 1 fully active ARV agent excluding NRTIs.
- Phase II Arm B: Phase I Then ENF 180mg QD: (Phase 1: ENF 90 mg SC BID): In the first phase or cohort phase of day I-1 through Week I-12 of the trial all patients received enfuvirtide (ENF) 90 mg subcutaneously (SC) twice daily (BID) + Isentress® [raltegravir] (RAL) 400-mg orally (PO) BID + optimized background (OB) with at least 1 fully active antiretroviral (ARV) agent excluding nucleoside reverse transcriptase inhibitor (NRTIs).
  In the randomized comparator phase Phase II of the trial- (Day II-1 through Week II-16): Virologic responders confirmed HIV-1 RNA ≤50 copies/mL)from Phase I were randomized to
  (Phase II Arm B: Phase I then ENF 180mg SC QD): ENF 180 mg SC once daily (QD) + RAL 400 mg PO BID + OB with at least 1 fully active ARV agent excluding NRTIs.
Arm/Group | Phase II Arm A: Phase I Then ENF 90mg BID | Phase II Arm B: Phase I Then ENF 180mg QD
Number analyzed (Participants) | 9 | 5
cells/mm3
  Phase I baseline to Week 1 of Phase II (n=8,5) | 22 [-39.0 to 139.0] | 118.0 [26.0 to 239.0]
  Phase I baseline to Week 12 of Phase II (n=7,4) | 83.0 [3.0 to 199.0] | 174.5 [-14.0 to 301.0]
  Phase I baseline to Week 16 of Phase II (n=6,4) | 61.0 [0.0 to 104.0] | 179.0 [18.0 to 225.0]

7. Secondary Outcome: Percentage of Patients With Ongoing Injection Site Reactions (ISRs)
Time Frame: Phase I and II
Measure: Number; unit: Percentage of patients
Groups:
- Phase II - Arm A: Phase I then ENF 90 mg SC BID
- Phase II - Arm B: Phase I then ENF 180 mg SC QD
Arm/Group | Phase I: ENF 90mg SC BID | Phase II - Arm A | Phase II - Arm B
Number analyzed (Participants) | 29 | 9 | 5
Percentage of patients
  Any type | 92 | 100 | 100
  Pain/discomfort | 52 | 42.9 | 60
  Erythema | 80 | 71.4 | 100
  Induration | 80 | 100 | 100
  Pruritus | 44 | 28.6 | 20
  Nodules | 56 | 57.1 | 80
  Ecchymosis | 40 | 14.3 | 20

ADVERSE EVENTS:
Time Frame: Phase I Day 1 through Week 12 & Phase II Day 1 through Week 16
Groups:
- Phase II Arm A: Phase I Then ENF 90mg SC BID: (Phase 1: ENF 90mg SC BID): In the first phase or cohort phase of day I-1 through Week I-12 of the trial all patients received enfuvirtide (ENF) 90 mg subcutaneously (SC) twice daily (BID) + Isentress® [raltegravir] (RAL) 400-mg orally (PO) BID + optimized background (OB) with at least 1 fully active antiretroviral (ARV) agent excluding nucleoside reverse transcriptase inhibitor (NRTIs).
  In the randomized comparator phase Phase II of the trial- (Day II-1 through Week II-16): Virologic responders confirmed HIV-1 RNA ≤50 copies/mL)from Phase I were randomized to
  (Phase II Arm A: Phase I then ENF 90mg SC BID): ENF 90 mg SC BID + RAL 400 mg PO BID + OB with at least 1 fully active ARV agent excluding NRTIs.
- Phase II Arm B: Phase I Then ENF 180mg SC QD: (Phase 1: ENF 90mg SC BID): In the first phase or cohort phase of day I-1 through Week I-12 of the trial all patients received enfuvirtide (ENF) 90 mg subcutaneously (SC) twice daily (BID) + Isentress® [raltegravir] (RAL) 400-mg orally (PO) BID + optimized background (OB) with at least 1 fully active antiretroviral (ARV) agent excluding nucleoside reverse transcriptase inhibitor (NRTIs).
  In the randomized comparator phase Phase II of the trial- (Day II-1 through Week II-16): Virologic responders confirmed HIV-1 RNA ≤50 copies/mL)from Phase I were randomized
  (Phase II Arm B: Phase I then ENF 180mg SC once daily (QD)): ENF 180 mg SC QD + RAL 400 mg PO BID + OB with at least 1 fully active ARV agent excluding NRTIs.
Arm/Group | Phase I: ENF 90mg SC BID | Phase II Arm A: Phase I Then ENF 90mg SC BID | Phase II Arm B: Phase I Then ENF 180mg SC QD
Serious Adverse Events (participants affected / at risk) | 4/29 | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 2/29 | 0/9 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: ENF 90mg SC BID (N=29) | Phase II Arm A: Phase I Then ENF 90mg SC BID (N=9) | Phase II Arm B: Phase I Then ENF 180mg SC QD (N=5)
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: ENF 90mg SC BID (N=29) | Phase II Arm A: Phase I Then ENF 90mg SC BID (N=9) | Phase II Arm B: Phase I Then ENF 180mg SC QD (N=5)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.